CLINICAL TRIAL: NCT02896166
Title: Microwave Ablation in the Treatment of Stage I Non Small Cell Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Xin Ye, Shandong Provincial Hospital affliated to Shandong University, Shandong Provincial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Shandong Provincial Hospital
Record Dates: First submitted 2016-08-20; First posted 2016-09-12 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Stage I NSCLC
Keywords: nsclc and stage I and microwave ablation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- microwave ablation (Experimental): The procedure is performed similar to a needle biopsy of the lung, under CT guidance. Placement of the needle-electrode is similar to needle placement for CT-guided biopsy. Appropriate positioning of the microwave ablation antenna is confirmed by CT imaging.
  Interventions: Other: microwave ablation

INTERVENTIONS:
Other: microwave ablation — eligible patients will be treated with microwave ablation in the primary tumor sites

SUMMARY:
Lung cancer, the leading cause of cancer related mortality. Among them, non small cell lung cancer accounts for 85%. Only part of patients could be treated with radical surgery, and some patients were unfit for surgery due to the poor cardio-pulmonary function or refuse surgery. For those patients, microwave ablation (MWA) could be an alternative treatment. Several small sample retrospective studies verified that MWA could be an efficacy and safe treatment.

DETAILED DESCRIPTION:
Patients with stage I non small cell lung cancer unfit for or refused surgery will be treated with MWA in the primary tumor sites.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has a histologically or cytologically verified NSCLC,
2. The tumors small enough to treat (usually <4 cm), and without chest pleura invasion.
3. Clinical stage I NSCLC with no other sites of disease,.
4. Patient is not a candidate for surgical removal of the cancer, or refused surgery.
5. Patient is not a candidate for radiation therapy, or refused radiation therapy.
6. Patient has > 6 month life expectancy.
7. Eastern Cooperative Oncology Group performance status of 0 to 2.
8. No prior anticancer treatments including surgery, radiation,chemotherapy or local treatments.
9. Sufficient organ functions.
10. Written informed consent.

Exclusion Criteria:

1. Active bacterial or fungous infection.
2. Simultaneous or metachronous (within the past 5 years) double cancers.
3. Women during pregnancy or breast-feeding.
4. Interstitial pneumonitis, pulmonary fibrosis, or severe pulmonary emphysema.
5. Uncontrollable diabetes mellitus.
6. History of severe heart disease, heart failure, myocardial infarction within the past 6 months or attack of angina pectoris within the past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From the date of randomization until the date of death from any cause，assessed up to 36 months

SECONDARY OUTCOMES:
Disease free survival | From the date of randomization until the date of first documented progression，assessed up to 36 months

OTHER OUTCOMES:
1-,2-, and 3-year survival rate | From the time of randomization to the end of 1-,2-, and 3-year,respectively

CONTACTS AND LOCATIONS:
Overall Officials: Xin Ye, M.D., Principal Investigator — Shandong Provincial Hospital affliated to Shandong University
Locations (2):
- China (2):
  - Shandong Provincial Hospital, Jinan, Shandong
  - Shandong Provincial Hospital affliated to Shandong University, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: No